CLINICAL TRIAL: NCT00556790
Title: Fast Track in Open Colonic Surgery - A Multicentric Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University of Zurich (Other); Kantonsspital Olten (Other); Kantonsspital Winterthur KSW (Other); Spital Uster (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 263/2003 USZ
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Elective Colectomie; Median Laparotomie
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Standard Care
  Interventions: Procedure: Standard Care
- 2 (Other): Fast Track Care
  Interventions: Procedure: Fast Track care

INTERVENTIONS:
Procedure: Standard Care — standard fluid regime, delayed feeding
  Arms: 1
Procedure: Fast Track care — restrictive fluid regime, early oral feeding, enforced mobilisation
  Arms: 2

SUMMARY:
To investigate the real value of a fast track protocol compared to a standard care protocol regarding postoperative complications and hospital stay in a multicentric setting in an intention to treat fashion.

DETAILED DESCRIPTION:
Our fast track protocol contains the four major components perioperative fluid restriction, epidural analgesia, early oral feeding and enforced mobilisation

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted for open colonic surgery

Exclusion Criteria:

* no primary anastomosis and/or stoma rectum resection emergency situation patients not speaking german immobile patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-11; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
complications until 30 days after surgery according to the zurich classification | 30 days postoperative

SECONDARY OUTCOMES:
hospital stay, adherence to Fast track protocol | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sven Muller, MD, Principal Investigator — University of Zurich
Locations (3):
- Switzerland (3):
  - Kantonsspital Olten, Olten
  - Spital Uster, Uster
  - Kantonsspital Winterthur, Winterthur

REFERENCES:
- [Derived] Hubner M, Muller S, Schafer M, Clavien PA, Demartines N. Impact of the nutritional risk score in fast-track colon surgery. Dig Surg. 2010;27(5):436-9. doi: 10.1159/000313692. Epub 2010 Nov 5. PMID 21051894
- [Derived] Muller S, Zalunardo MP, Hubner M, Clavien PA, Demartines N; Zurich Fast Track Study Group. A fast-track program reduces complications and length of hospital stay after open colonic surgery. Gastroenterology. 2009 Mar;136(3):842-7. doi: 10.1053/j.gastro.2008.10.030. Epub 2008 Nov 1. PMID 19135997